CLINICAL TRIAL: NCT05994352
Title: The Effect Of Vırtual Realıty Applıcatıon On Therapeutıc Communıcatıon Skılls Levels Of Mental Health And Psychıatrıc Nursıng Students
Brief Title: Psychiatric Nursing Students Therapeutic Communication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Arzu Dikici, lecturer, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IstanbulArelU
Record Dates: First submitted 2023-07-12; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Communication
Keywords: therapeutic; communication; mental health; nursing; student
MeSH Terms: conditions — Communication; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): no intervention will be applied to the students in the control group
- experimental group (Experimental): virtual reality simulation will be applied to the experimental group
  Interventions: Other: virtual reality simulation

INTERVENTIONS:
Other: virtual reality simulation — The effect of virtual reality simulation on therapeutic communication skill levels
  Arms: experimental group

SUMMARY:
This research was carried out to determine the effect of virtual reality application on the therapeutic communication skill levels of Mental Health and Psychiatric Nursing course students. The research was carried out in experimental research design. The independent variable of the research is virtual reality simulation; The dependent variable is the therapeutic communication skills of the students of the Mental Health and Psychiatric Nursing course. Nursing students' individual characteristics were determined as the control variable. The hypothesis of the research H1: The therapeutic communication skill level scores of the nursing students in the intervention group participating in the virtual reality simulation will increase compared to the nursing students in the control group.

DETAILED DESCRIPTION:
This research was carried out to determine the effect of virtual reality application on the therapeutic communication skill levels of Mental Health and Psychiatric Nursing course students. The analysis was carried out in an experimental research design. The independent variable of the study is virtual reality simulation; The dependent variable is the therapeutic communication skills of the students of the Mental Health and Psychiatric Nursing course. Nursing students' characteristics were determined as the control variable. The hypothesis of the research H1: The therapeutic communication skill level scores of the nursing students in the intervention group participating in the virtual reality simulation will increase compared to those in the control group. The population of the research consists of 65 students who are enrolled in the nursing department of a foundation university in Istanbul and took the mental health and psychiatric nursing course in the spring term of the 2022-2023 academic year. Sample: A list from 1 to 65 was prepared to determine the students who will take place in the intervention and control groups. Simple random sampling method was used to differentiate between intervention and control groups. The numbers to be sampled were determined by www.random.org generate number. The intervention group consisted of 36 students and the control group consisted of 29 students.

ELIGIBILITY:
Inclusion Criteria:

* • To be registered in the Mental Health and Psychiatric Nursing course in the spring semester of the 2022-2023 academic year,

  * To be taking the Mental Health and Psychiatric Nursing course for the first time in the nursing department,
  * To attend school regularly,
  * Not having received training with virtual reality simulation within the scope of Mental Health and Psychiatric Nursing course.

Exclusion Criteria:

-

Ages: 20 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The therapeutic communication skill levels of mental health and psychiatric nursing students | 4 mounth
  descriptive characteristics of the participants. The form, consisting of 7 questions in total, containing information such as the age, gender, place of residence of the students for the longest time, presence of mental illness, was prepared by the researcher using the literature
Nursing students' therapeutic communication skills | 4 mounth
  The scale developed by Karaca, et al. (2019) was designed as a measurement tool for determining the therapeutic communication skills of nursing students. The scale consists of 16 items and 3 sub-dimensions: "Non-therapeutic Communication Skills", "Therapeutic Communication Skills-1", "Therapeutic Communication Skills-2". The first sub-dimension of my scale consists of 7 items, the second sub-dimension consists of 6 items and the third sub-dimension consists of 3 items. The scale is 7-point Likert type varying between 1 and 7, there is no reverse coded item in the scale. The highest score that can be obtained from the scale is 16x7=112, and the lowest score is 16x1=16.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Dikici, Principal Investigator — lecturer
Locations (1):
- Istanbul Arel University, Istanbul, Turkey (Türkiye)